CLINICAL TRIAL: NCT03364010
Title: Relationships Between Proprioception, Motor Control and Reading in Children With Dyslexia
Brief Title: Dyslexia, Motor Control and Proprioception
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: END OF INCLUSIONS
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C17-14; 2017-A01547-46 (Registry Identifier: RCB)
Record Dates: First submitted 2017-09-27; First posted 2017-12-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Dyslexia
Keywords: Motor control; Proprioception
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dyslexic and non dyslexic Children (Experimental): Children aged 10-12 Evaluation of proprioception Evaluation of motor learning Evaluation of written language
  Interventions: Behavioral: Evaluation of proprioception; Behavioral: Evaluation of motor learning; Behavioral: Evaluation of written language

INTERVENTIONS:
Behavioral: Evaluation of proprioception — Velocity perception and Position perception
Behavioral: Evaluation of motor learning — Motor accurancy and State Estimation with visual perturbations
Behavioral: Evaluation of written language — Text reading, Identifying words and Phonological awareness: phonemic blending and phonemic elision

SUMMARY:
The investigators hypothesize that children with dyslexia present proprioceptive disorders and the purpose of the present study is to better understand relationships between motor control, proprioception and academic learnings. The investigators compare a group of French students with and without dyslexia aged 10-12.

DETAILED DESCRIPTION:
2 groups of children (dyslexics and control) will be evaluated on 2 tasks:

* Evaluation of the proprioception: Perception of the speed and Perception of the position
* Evaluation of the motor learning: Estimation of state in the framework of a motor perturbation

ELIGIBILITY:
Inclusion criteria for all children

* Child with a French social security
* School child
* Native French speaker
* right-handed
* Normal or corrected vision
* Without neurological or psychiatric histories
* Agree to participate in the study in agreement with parental rights representatives

For the dyslexic group :

* pluridisciplinary diagnostic
* never consulted for proprioception before
* without any other leaning disorders like dysphasia
* attention deficit hyperactivity disorder (ADHD) or developmental coordination disorder (DCD)

For the control group :

* regular school attendance
* never consulted for learning disabilities
* No learning disorders known for their parents or siblings.

Exclusion criteria for all children

* genetic disorder
* neurological or psychiatric history
* Delayed psychomotor development
* Reeducation or current treatment interfering with the evaluation

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of proprioception through velocity perception | 1day
  The ability to perceive motion at 3 different velocities for 3 different joints is assessed using a motorized ergometer. A passive movement is performed by the ergometer and children are tasked to press a button as soon as they feel the movement. We calculate the angle of detection for each speed and compare it between Dyslexic and healthy children.

SECONDARY OUTCOMES:
Evaluation of proprioception through position perception | 1 day
  The ability to perceive position is assessed using an ergometer that produces passive movements of 3 different amplitudes on the dominant arm. In a second time, the ergometer produces a passive movement of the same arm and children are tasked to press a button as soon as they feel they are in the exact previously-experienced position. We calculate the angular error and compare it between Dyslexic and healthy children.
Motor learning | 1 day
  The ability to learn new motor tasks is assessed using virtual reality and motor acquisition systems. First we evaluate the motor accuracy and the state estimation by pointing tests. Then visual perturbations are introduced during pointing. Finally, we evaluate motor accuracy and state estimation again.
Text reading | 1day
  The ability to read aloud a text is assessed using the French standardized test " Alouette ", which provide accuracy in reading aloud age-normed texts (ratio between words that have been correctly read and all the words that have been read).
Phonological awareness: phonemic blending and phonemic elision | 1day
  The ability to derive a phonemic pattern from distinct phonemic units or to substitute a phonemic pattern for another is assessed using the French standardized test " Nepsy2, phonological process " which provide standard deviation in reading aloud by the investigator.
Identifying words | 1day
  The ability to identify words is assessed using the French standardized test " Timé3 ", which provide lexical level and delay reading in silent reading age-normed words.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick QUERCIA, dr, Principal Investigator — Unité Inserm d'affiliation : Laboratoire U1093 Cognition, Action et Plasticité Sensorimotrice
Locations (1):
- Inserm U1093, Dijon, Bourgogne-Franche-Comté, France

REFERENCES:
- [Derived] Laprevotte J, Papaxanthis C, Saltarelli S, Quercia P, Gaveau J. Movement detection thresholds reveal proprioceptive impairments in developmental dyslexia. Sci Rep. 2021 Jan 11;11(1):299. doi: 10.1038/s41598-020-79612-4. PMID 33431949